CLINICAL TRIAL: NCT01166672
Title: Weight Loss to Prevent BCRL: A Pilot Study
Brief Title: BCRL Prevention Pilot
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15110
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Breast Cancer
Keywords: obese women (BMI greater than or equal to 30), do not already have a diagnosis of lymphedema, who are done; with surgery, chemotherapy, and radiation therapy, and who were diagnosed with breast cancer within the; past 2 years will be invited to participate.
MeSH Terms: conditions — Obesity; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to establish feasiblity of recruiting obese breast cancer survivors at the end of treatment, getting those survivors to lose weight and attend follow-up visits for 6 months.

DETAILED DESCRIPTION:
Breast cancer related lymphedema occurs in 20-30% of survivors. Weight loss could prevent onset. We seek to do a pilot study to establish feasibility of 1) recruiting survivors at risk for lymphedema to do a weight loss intervention, 2) achieving 10-15% weight loss over 26 weeks in this population, and 3) attendance at follow-up visits 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Breast Cancer Survivors who had 5 or more lymph nodes removed and radiation to lymph nodes as part of treatment.
* Completed all treatments - no metastatic cancers
* Overweight or obese (BMI greater than or equal to 25 kg/m2)
* Medically and logistically able to participate in a weight loss and exercise program over 6 months.
* Diagnosed with breast cancer within the past 2 years.

Exclusion Criteria:

* More than 2 years since breast cancer diagnosis
* Medical status that would preclude safety of participation in a weight loss and exercise program
* Metastatic cancer
* Already enrolled in a weight loss program

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, aged 18-70, who are obese (BMI greater than or equal to 30), do not already have a diagnosis of lymphedema, who are done with surgery, chemotherapy, and radiation therapy, and who were diagnosed with breast cancer within the past 2 years will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Follow-up Appts. | 6 months
  The primary outcome will be the precent of participants who complete 6 month follow-up appointments.

SECONDARY OUTCOMES:
Response Rates | 6 months
  Secondary outcomes will include response rates (% approached who enroll, consent, and attend intervention sessions), weight loss at 6 months, and arm volumes and lymphedema survey responses at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States